CLINICAL TRIAL: NCT02447666
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Activity of Azacitidine and to Compare Azacitidine to Historical Controls in Pediatric Subjects With Newly Diagnosed Advanced Myelodysplastic Syndrome or Juvenile Myelomonocytic Leukemia Before Hematopoietic Stem Cell Transplantation
Brief Title: Study With Azacitidine in Pediatric Subjects With Newly Diagnosed Advanced Myelodysplastic Syndrome (MDS) and Juvenile Myelomonocytic Leukemia (JMML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-JMML-001
Record Dates: First submitted 2015-04-14; First posted 2015-05-19 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Myelodysplastic Syndrome; Leukemia, Myelomonocytic, Juvenile
Keywords: Azacitidine; Myelodysplastic syndrome; Juvenile myelomonocytic leukemia; Hematopoietic stem cell transplantation; Vidaza; Hypomethylating agent
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine Myelodysplastic Syndrome (MDS) (Experimental): Azacitidine 75 mg/m2 by Intravenous (IV) or Subcutaneous (SC) administration once daily (QD) on Days 1 to 7 of a 28-day cycle for a minimum of 3 cycles and a maximum of 6 cycles.
  Interventions: Drug: Azacitidine
- Azacitidine Juvenile Myelomonocytic Leukemia (JMML) (Experimental): Azacitidine 75 mg/m2 by Intravenous (IV) or Subcutaneous (SC) administration once daily (QD) on Days 1 to 7 of a 28-day cycle for a minimum of 3 cycles and a maximum of 6 cycles.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine
  Other Names: Vidaza

SUMMARY:
Indication Treatment of pediatric subjects with newly diagnosed advanced myelodysplastic syndrome (MDS) or juvenile myelomonocytic leukemia (JMML) prior to hematopoietic stem cell transplantation (HSCT).

Objectives Primary Objective The primary objective is to assess the treatment effect on response rate (MDS: either complete remission [CR], partial remission [PR], or marrow CR; JMML: either clinical complete remission [cCR] or clinical partial remission [cPR]); at Cycle 3 Day 28 (each cycle is 28 days) and to compare against standard therapy using a matched-pairs analysis of historical data.

Secondary Objective The secondary objective is to further evaluate safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of azacitidine in this subject population.

Study Design This is a prospective, open-label, Phase 2 study consisting of 2 parallel experimental arms, one for each disease group: MDS and JMML. Each arm is designed based on Simon's Optimal 2 stage study design. The sample size has been calculated to allow evaluation of the response rate at 28 day-Cycle 3 Day 28 in each of the 2 disease groups. Each of the experimental arms will also individually be compared against a historical control arm using data retrospectively collected from the European Working Group of MDS in childhood (EWOG-MDS) registry by means of a matched-pairs analysis; matched for predefined subject baseline characteristics defined before any results from this study are known post Stage 1. If matched pair is not viable then other methodologies will be explored to evaluate and compare response rates reported in literature and also in registry database Twenty subjects with MDS and 35 JMML subjects evaluable for the primary endpoint (ie, subjects that receive at least 1 dose of investigational product [IP]) will be enrolled at approximately 45 centers in Europe. Each experimental arm has 1 interim analysis planned (at the end of Stage 1). If, during Stage 1 evaluation, less than 2 subjects are observed with a CR, PR, or marrow CR after 3 months of azacitidine in the first 9 subjects with MDS, then enrollment will be stopped. Similarly, if less than 3 subjects are observed with a cPR or cCR after 3 months of azacitidine in the first 18 subjects with JMML, then enrollment will be stopped.

DETAILED DESCRIPTION:
Study Population Pediatric subjects aged 1 month to less than 18 years of age with newly diagnosed conditions of advanced myelodysplastic syndrome (MDS) or juvenile myelomonocytic leukemia (JMML).

Length of Study The enrollment period will last for up to 22 months with subjects being treated for a minimum of 3 months and a maximum of 6 months, until transplantation or disease progression (based on an independent central review of responses). Once investigational product (IP) has been discontinued, subjects will then be followed for 1 year after the last dose of investigational product (IP). The follow-up may not be terminated because of new anticancer treatment or hematopoietic stem cell transplantation (HSCT).

The End of Trial is defined as either the date of the last visit of the last subject to complete the study, or the date of receipt of the last data point from the last subject that is required for primary, secondary and/or exploratory analysis, as pre-specified in the protocol and/or the Statistical Analysis Plan (SAP), whichever is the later date.

ELIGIBILITY:
Inclusion Criteria:

Myelodysplastic Syndromes (MDS) :

1. Understand and voluntarily provide permission (subjects and/or when applicable, parental/legal representative) to the informed consent form/informed assent form (ICF/IAF) prior to conducting any study-related assessments/procedures.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Male or female age 1 month to less than 18 years old at the time of informed consent/informed assent.
4. Newly diagnosed advanced primary or secondary Myelodysplastic Syndromes (MDS), with latest peripheral blood (PB) and bone marrow (BM) biopsy confirming diagnosis within the 14 days prior to informed consent signature, with one of the following:

   1. RAEB (Refractory anemia with excess blasts): 2% to 19% blasts in PB or 5% to 19% blasts in BM.
   2. RAEB-t (Refractory anemia with excess blasts in transformation): 20% to 29% of blasts in PB or BM.
   3. Secondary Myelodysplastic Syndromes presenting as chronic myelomonocytic leukemia (CMML) without increase in blasts but with chromosomal abnormality
5. Lansky play score at least equal to 60; or Karnofsky performance status at least equal to 60.
6. Life expectancy of at least 3 months.
7. Normal renal function defined as less than or equal to NCI CTCAE (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]) v 4.0 Grade 1 (maximum 1.5 x Upper Limit of Normal [ULN]).
8. Normal liver function defined as less than or equal to NCI CTCAE v 4.0 Grade 1 (maximum 2.5 x ULN for transaminases and bilirubin).
9. Females of childbearing potential and male subjects that have reached puberty and are younger than 18 years of age must agree to undergo physician-approved reproductive education and discuss the side effects of the Investigational Product (IP) on reproduction with parent(s) and/or guardian(s).
10. Females of childbearing potential, defined as females who have achieved menarche and/or 8 years or older and have not undergone a hysterectomy or bilateral oophorectomy, must meet the following conditions below. (Note: Amenorrhea following cancer therapy does not rule out childbearing potential):

    1. Have a negative serum pregnancy test within 72 hours prior to starting IP as verified by the Investigator. Agree to ongoing pregnancy testing during the course of the study
    2. Female subjects must, as appropriate to age and the discretion of the study physician, either commit to true abstinence1 from heterosexual contact (which must be reviewed on a monthly basis) and/or agree to the use of approved contraceptive method (eg. oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; or vasectomized partner) while on azacitidine; and for 3 months following the last dose.
11. Male subjects must, as appropriate to age and the discretion of the study physician:

    1. Agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential (FCBP) while participating in the study, during dose interruptions, and for at least 3 months following azacitidine discontinuation, even if he has undergone a successful vasectomy.

Juvenile Myelomonocytic Leukemia Subjects (JMML):

1. Understand and voluntarily provide permission (subjects and/or when applicable, parental/legal representative) to the ICF/IAF prior to conducting any study-related assessments/procedures.
2. Able to adhere to the study visit schedule and other protocol requirements.
3. Male or female age 1 month to less than 18 years old at the time of informed consent/informed assent.
4. Newly diagnosed Juvenile Myelomonocytic Leukemia (JMML), with PB and BM confirming diagnosis prior to informed consent signature, with one of the following

   1. somatic mutation in PTPN11
   2. somatic mutation in KRAS
   3. somatic mutation in NRAS and HbF % > 5x normal value for age
   4. clinical diagnosis of neurofibromatosis Type 1.
5. Lansky play score at least equal to 60; or Karnofsky performance status at least equal to 60.
6. Life expectancy of at least 3 months.
7. Normal renal function defined as less than or equal to NCI CTCAE v 4.0 Grade 1 (maximum 1.5 x ULN).
8. Normal liver function defined as less than or equal to NCI CTCAE v 4.0 Grade 1 (maximum 2.5 x ULN for transaminases and bilirubin).
9. Females of childbearing potential and male subjects that have reached puberty and are younger than 18 years of age must agree to undergo physician-approved reproductive education and discuss the side effects of the IP on reproduction with parent(s) and/or guardian(s).
10. Females of childbearing potential, defined as females who have achieved menarche and/or 8 years or older and have not undergone a hysterectomy or bilateral oophorectomy, must meet the following conditions below.

    1. Have a negative serum pregnancy test within 72 hours prior to starting IP as verified by the Investigator. Agree to ongoing pregnancy testing during the course of the study
    2. Female subjects must, as appropriate to age and the discretion of the study physician, either commit to true abstinence2 from heterosexual contact (which must be reviewed on a monthly basis) and/or agree to the use of approved contraceptive method (eg. oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; or vasectomized partner) while on azacitidine; and for 3 months following the last dose.
11. Male subjects must, as appropriate to age and the discretion of the study physician:

    a. Agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential (FCBP) while participating in the study, during dose interruptions, and for at least 3 months following azacitidine discontinuation, even if he has undergone a successful vasectomy.
12. SO2 greater than 92% (without additional supply of O2).
13. Peripheral blood monocyte count of at least 1.0 x 109/L.
14. Blast percentage in PB and BM less than 20%.
15. Splenomegaly.

Exclusion Criteria:

Myelodysplastic Syndromes (MDS):

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Treated by any investigational agent in a clinical study within 4 weeks prior to signing of informed consent / informed assent.
5. Any central nervous system (CNS) involvement.
6. Isolated extramedullary disease.
7. Current uncontrolled infection.
8. Cardiac toxicity (shortening fraction below 28%).
9. Concurrent treatment with another anticancer therapy.
10. Pregnancy or lactation.
11. Prior treatment with a demethylating agent.
12. Allergy to azacitidine or mannitol.
13. Any other organ dysfunction (NCI-CTCAE v 4.0 Grade 4) that will interfere with the administration of the therapy according to this protocol.
14. Genetic abnormalities indicative of Core Binding factor AML; t(8;21), inv16, t(16;16), and t(15;17).
15. Subjects with inherited BM failure syndromes (ie, Fanconi's anemia, congenital severe neutropenia, Shwachman-Diamond syndrome).

Juvenile Myelomonocytic Leukemia Subjects:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Treated by any investigational agent in a clinical study within 4 weeks prior to signing of informed consent / informed assent.
5. Any CNS involvement.
6. Isolated extramedullary disease.
7. Current uncontrolled infection.
8. Cardiac toxicity (shortening fraction below 28%).
9. Concurrent treatment with another anticancer therapy.
10. Pregnancy or lactation.
11. Prior treatment with a demethylating agent.
12. Allergy to azacitidine or mannitol.
13. Any other organ dysfunction (NCI-CTCAE v 4.0 Grade 4) that will interfere with the administration of the therapy according to this protocol.
14. Germline molecular aberrations in CBL, PTPN11, NRAS, or KRAS.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Myelodysplastic Syndrome (MDS) response rate at end of third 28-day cycle | Up to 4 Months
  Defined as proportion of subjects with complete remission [CR], partial remission [PR] or marrow CR according to modified criteria described by Cheson 2006, adapted to pediatric reference values at 3 months (28 days cycle). Response must be sustained for at least 4 weeks either in the 4-week period preceding or succeeding 3 months (ie, sustained over the period minimum 2 months to end of 3 months, or end of 3 months to end of 4th months).
Juvenile Myelomonocytic Leukemia (JMML) response rate at end of 3 Months | Up to 4 Months
  Defined as proportion of subjects with sustained clinical complete remission [cCR] or clinical partial remission [cPR] according to the International JMML response criteria in Niemeyer 2014 at 3 months (28 days cycles). Response must be sustained for at least 4 weeks either in the 4-week period preceding or succeeding 3 months (ie, sustained over the period minimum 2 months to end of 3 months, or end of 3 monthsto end of 4 months).

SECONDARY OUTCOMES:
Cytogenetic response for MDS | Up to 6 Months
  Cytogenetic response is defined as the number of subjects with complete disappearance of the chromosomal abnormality without appearance of new ones divided by the number of subjects within the analysis population.
Cytogenetic response for JMML subjects | Up to 6 Months
  Cytogenetic response is defined as the number of subjects with complete disappearance of the chromosomal abnormality without appearance of new ones divided by the number of subjects within the analysis population.
Molecular Response for JMML subjects | Up to 6 Months
  Molecular response is defined as the number of subjects with absence of somatic mutations related to JMML divided by the number of subjects within the analysis population.
Duration of Response (CR, PR or marrow CR) for MDS patients | Up to 30 months
  Duration of response will consist of only the subjects achieving a response (CR, PR or marrow CR) and is defined as the time from first observed response until either disease progression or any cause of death.
Duration of Response (Clinical CR or Clinical PR) for JMML patients | Up to 18 months
  Duration of response will consist of only the subjects achieving a response (cCR or cPR) and is defined as the time from first observed response until either disease progression or any cause of death.
Time to Response (TTR) for MDS patients | Up to 6 Months
  TTR is defined as the time from first study dose day until a response of CR, PR or marrow CR, whichever occurs first. Only subjects observed with a response will be included in the analysis with the median TTR across the subjects presented.
TTR of Clinical CR or Clinical PR for JMML patients | Up to 6 Months
  Time to Response (TTR) is defined as the time from first study dose day until a response cCR or cPR, whichever occurs first. Only subjects observed with a response will be included in the analysis with the median TTR across the subjects presented.
Time to Progression (TTP) | Up to 18 months
  Time to Progression (TTP) is defined as the time from first study dose day until either disease progression or death due to progression.
Leukemia free survival (LFS) | Up to 18 months
  Leukemia free survival (LFS) is defined as the time from HEMATOPOIETIC STEM CELL transplant (HSCT) date until leukemia progression or death for subjects receiving a HSCT only. Subjects alive and leukemia-free at the time of the statistical analysis will be censored at the time of their last disease assessment. Subjects will also be censored at the time of starting a new anticancer therapy if having not previously had a leukemia progression.
Overall survival (OS) | Up to 18 months
  OS is defined as the time from first study dose day until death from any cause. Subjects alive at the time of analysis will be censored at the time they were last known to be alive.
Deoxyribonucleic acid methylation status in (BM) | Up to 18 months
  DNA methylation levels will be assessed across time points by means of a repeated measures analysis of variance (ANOVA) test thereby allowing identification of possible changes in methylation levels over time by treatment arm as well as comparing DNA methylation levels between treatment arms per disease indication
Percentage of subjects undergoing HSCT | Up to 18 months
  Defined as the proportion of subjects undergoing HSCT during the conduct of this study over the total number of subjects enrolled into this study.
Time to first HSCT | Up to 18 months
  The time from first study dose day until HSCT date. Subjects not receiving a HSCT will be censored at the time of the analysis.
Adverse Events (AEs) | Up to 7 months
  All reported adverse events during the duration of the study conduct.
Pharmacokinetic parameters of azacitidine; Cmax | Up to 28 days
  Cmax is defined as the observed maximum plasma concentration
Pharmacokinetic parameters of azacitidine; Tmax | Up to 28 days
  Tmax is defined as the observed time to maximum plasma concentration
Pharmacokinetic parameters of azacitidine; AUCt | Up to 28 days
  Area under the plasma concentration-time curve from time zero to the last quantifiable time point
Pharmacokinetic parameters of azacitidine; area under the plasma concentration-time curve from time zero to infinity (AUC ∞) | Up to 28 days
  The AUC ∞ is defined as area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetic parameters of azacitidine; Terminal Rate λz | Up to 28 days
  Terminal phase rate constant is determined by linear regression of the terminal points of the log-linear plasma concentration-time curve
Pharmacokinetic parameters of azacitidine; terminal phase half-life | Up to 28 days
  The Terminal phase half-life will be calculated according to the following equation: t½ = 0.693/λz
Pharmacokinetic parameters of azacitidine; total clearance (CL) | Up to 28 days
  The total clearance is calculated as Dose/AUC∞
Pharmacokinetic parameters of azacitidine; volume of distribution (Vz) | Up to 28 days
  The volume of distribution will be calculated according to the equation: Vz = (CL)/λz

CONTACTS AND LOCATIONS:
Overall Officials: Bouchra Benettaib, MD, Study Director — Celgene Corporation
Locations (39):
- St. Anna Kinderkrebsforschung, CHILDREN'S CANCER RESEARCH INSTITUTE, Vienna, Austria
- Belgium (2):
  - Hopital Universitaire des Enfants, Brussels
  - University Hospital Ghent, Ghent
- University Hospital Motol, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Centre Hospitalier Universitaire Lyon, Lyon
  - Hopital d'Enfants de la Timone, Marseille
  - Hopital Robert Debre, Paris
- Germany (15):
  - Klinikum Augsburg, Augsburg
  - Charite Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Hematology, Oncology and clinical immunology / Heinrich-Heine-University, Düsseldorf
  - Universitatsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt/Main, Frankfurt am Main
  - Universitatsklinik, Freiburg im Breisgau
  - University of Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum, Jena
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Klinikum der Universitaet Muenchen, München
  - Universitatsklinik Munster, Münster
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Universitatsklinikum, Tübingen
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- Italy (7):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - IRCCS Gaslini Hospital, Genova Quarto
  - Azienda Ospedaliera San Gerardo, Monza
  - General Hospital, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale Bambin Gesu, Roma
  - Regina Margherita Children's Hospital, Torino
- Erasmus University Medical Center, Rotterdam, Netherlands
- Spain (3):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Virgen de La Arrixaca, Murcia
- Sweden (2):
  - Queen Silvia Childrens Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
- Universitäts-Kinderklinik, Zurich, Switzerland
- Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Niemeyer CM, Flotho C, Lipka DB, Stary J, Rossig C, Baruchel A, Klingebiel T, Micalizzi C, Michel G, Nysom K, Rives S, Schmugge Liner M, Zecca M, Schonung M, Baumann I, Nollke P, Benettaib B, Biserna N, Poon J, Simcock M, Patturajan M, Menezes D, Gaudy A, van den Heuvel-Eibrink MM, Locatelli F. Response to upfront azacitidine in juvenile myelomonocytic leukemia in the AZA-JMML-001 trial. Blood Adv. 2021 Jul 27;5(14):2901-2908. doi: 10.1182/bloodadvances.2020004144. PMID 34297046
- See also: Expanded Access for CC-486 — https://clinicaltrials.gov/ct2/show/NCT02447666?term=AZA-JMML-001&rank=1